CLINICAL TRIAL: NCT05253391
Title: Adequacy of Management of Patients With Asthma Exacerbation in Martinique
Acronym: APEXA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 20_RIPH3-18
Record Dates: First submitted 2022-01-28; First posted 2022-02-23 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Asthma
Keywords: Asthma; Asthma exacerbation; Acute asthma; Emergency; Asthma treatment; French West Indies
MeSH Terms: conditions — Asthma; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated for asthma exacerbation
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Routine care — The investigator takes care of the patient according to the protocol in force in his department and decides on the final orientation of the patient (transfer to intensive care unit/ICU, hospitalization or home discharge).
  No recommendations or instructions are given to the investigators. Each investigator is free to decide on his care and the terms of transfer, hospitalization and discharge.

SUMMARY:
Asthma is a chronic respiratory disease whose goal of therapeutic, educational and preventive care is to prevent the onset of acute crisis, the most serious of which are life threatening. A general population survey shows a greater prevalence of asthma in the French West Indies compared to hexagonal France, but there is no data to our knowledge on asthma exacerbations requiring pre and intra-hospital emergency services, nor on the clinical severity or on the adequacy of the therapeutic care.

Asthma exacerbations, in particular serious forms requiring immediate admission to the Emergency Department or Intensive Care Unit or leading to hospitalization, can be considered as a failure in the prevention of crisis and therefore disease control. The management of acute or subacute asthma exacerbations is however well codified in expert recommendations, renewed annually by the Global Initiative for Asthma (GINA). These recommendations specify not only the initial care, but also the strategy and modalities of return home and post-emergency follow-up. Recently the French Language Resuscitation Society (SRLF) and the French Society of Emergency Medicine (SFMU) jointly published formalized expert recommendations (RFE) on the management of asthma exacerbations (Le Conte 2019).

These RFEs still remain the benchmark in France for adequate management of asthma exacerbations for adults and children. Despite these updated recommendations, field observations often show inadequate care, both in the emergency and in the post-emergency period.

DETAILED DESCRIPTION:
The rationale for this study is based on the lack of data concerning the characteristics of asthma exacerbations and their emergency management in Martinique, but also the lack of awareness of the adequacy of this management according to the stage of severity, as recommended.

Better knowledge of asthma exacerbations, of the stage of clinical severity, of emergency treatments and of post-emergency follow-up, would improve the overall care of asthma patients in Martinique and induce a better control their disease.

This prospective clinical research includes all the services of the Martinique University Hospital which take care of asthma patients during or after their exacerbation: Emergency medical assistance service (SAMU), Mobile emergency and resuscitation structure (SMUR), adult and pediatric emergency services, adult and pediatric resuscitation and pulmonology service.

In order not to guide or influence the therapeutic decisions of the investigators in charge of the patients in this study, and because the evaluation of the adequacy of the management according to the stage of severity is the main objective of the study, no recommendations or instructions are given to the investigators. Each investigator freely decides on the treatment (diagnosis, assessment of severity, treatment, modalities and prescription for discharge from emergencies, hospitalization or not).

This research is the first assessment of asthma exacerbations carried out in our region with the aim of improving their management in order to limit their prognostic impact.

ELIGIBILITY:
Inclusion Criteria:

* All children and adolescents (2-17 years) and adults (≥ 18 years) asthma patients.
* Supported either by a team from mobile emergency and resuscitation service (SMUR) participating in the study, or by a team from the Emergency Department or possibly admitted directly to an intensive care unit participating in the study.
* With an asthma exacerbation (acute asthma), the diagnostic criteria of which are as follows: history of asthma or wheezing dyspnea, exacerbation of wheezing, difficulty breathing, shortness of breath, wheezing or dry cough, and finally wheezing or silence on auscultation.
* Patient or patient representative who has given oral consent for the use of their medical data for this research.

Exclusion Criteria:

* Patient with a strong suspicion or a proven diagnosis of acute respiratory failure on chronic respiratory failure.
* Patient with a strong suspicion or a proven diagnosis of acute left heart failure with wheezing (cardiac asthma) or crackling rales.
* Patient with a strong suspicion or a proven diagnosis of acute febrile pneumonitis.
* Patient with a strong suspicion or a proven diagnosis of acute pleurisy (reduction or elimination of vesicular murmurs, dullness of the bases or imaging).
* Patient or representative of the patient who refused to agree to his participation in the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated for asthma exacerbation.
Sampling Method: Non-Probability Sample
Enrollment: 339 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
To assess the adequacy of the management of acute asthma exacerbations according to the stage of severity for patients treated at the CHU of Martinique. | 19 months
  Percentage of patients who received adequate management by stage of severity of acute exacerbation. A tool to assist in the management of an exacerbation of asthma is described to define adequate or non-adequate management by an expert committee.

SECONDARY OUTCOMES:
Describe the distribution of the different stages of severity of asthma exacerbations. | 19 months
  Percentage of each of the 3 severity stages of acute asthma exacerbations.
Measure the hospitalization rate according to the stage of severity of the asthma exacerbations. | 19 months
  Hospitalization rate (emergency unit, intensive care unit or medical or pneumology department) according to the initial stage of severity.
Measure the rate of recurrence of exacerbation (for SAMU, Emergencies, resuscitation or hospitalization) within 30 days of the initial crisis. | 19 months
  Acute exacerbation recurrence rate (SAMU, Emergency, resuscitation or hospitalization) within 30 days of the first inclusion.
Measure the incidence during the study period of asthma exacerbations treated urgently at the CHU of Martinique. | 19 months
  Incidence rate of acute exacerbations during the study period.
Measure the proportion of patients having an exit treatment including a background treatment. | 19 months
  Proportion of patients having an exit treatment including a background treatment.
Measure the proportion of patients who actually took their background treatment at day 30 after the crisis. | 30 days
  Proportion of patients who actually took their background treatment at day 30 after the crisis.

CONTACTS AND LOCATIONS:
Locations (7):
- Martinique (7):
  - CHU of Martinique - Emergency Department of Pierre Zobda Quitman, Fort-de-France
  - CHU of Martinique - Pediatric Emergency Unit, Fort-de-France
  - CHU of Martinique - Pediatric Resuscitation Unit, Fort-de-France
  - CHU of Martinique - Pneumology Service, Fort-de-France
  - CHU of Martinique - Resuscitation Unit, Fort-de-France
  - CHU of Martinique - SAMU/SMUR, Fort-de-France
  - CHU of Martinique - Emergency Department of Trinité, La Trinité

IPD SHARING:
Plan to Share IPD: No